CLINICAL TRIAL: NCT03711851
Title: Managing Chronic Pain Through Self-Help: A Randomized Controlled Trial Comparing Guided Self-Help Programs Based on Acceptance and Commitment Therapy (ACT) to Education
Brief Title: Managing Chronic Pain Through Self-Help
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Quebec Pain Research Network (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Dr. Frédérick Dionne, Ph.D., Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDERS-17-11-06.05
Record Dates: First submitted 2018-10-09; First posted 2018-10-19 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Self-help; Bibliotherapy; Web-based interventions; Acceptance and commitment therapy; Psychological flexibility
MeSH Terms: conditions — Chronic Pain | interventions — Bibliotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web-based (Experimental): Self-help Acceptance and commitment therapy (Web-based)
  Interventions: Behavioral: Self-help Acceptance and commitment therapy (Web-based)
- Bibliotherapy (Experimental): Self-help Acceptance and commitment therapy (bibliotherapy)
  Interventions: Behavioral: Self-help Acceptance and commitment therapy (bibliotherapy)
- Education pamphlets on pain (Active Comparator): Self-help Education on Chronic pain (pamphlet style pdf documents)
  Interventions: Other: Self-help Education pamphlets on pain (active control group)

INTERVENTIONS:
Behavioral: Self-help Acceptance and commitment therapy (Web-based) — 9 week program with minimal contact with therapist (predominantly self-help)
  Arms: Web-based
Behavioral: Self-help Acceptance and commitment therapy (bibliotherapy) — 9 week program with contact with therapist (predominantly self-help)
  Arms: Bibliotherapy
Other: Self-help Education pamphlets on pain (active control group) — 9 week program with contact with therapist (predominantly self-help)
  Arms: Education pamphlets on pain

SUMMARY:
Chronic pain has a significant impact on the physical and emotional functioning of those living with this condition. It is now recognized that Acceptance and Commitment Therapy (ACT) is an effective treatment in managing chronic pain; however, several barriers limit its accessibility. Therefore, self-help versions of ACT are promising because they offer a cost-effective treatment option that usually require little support from a therapist, and can be widely accessed.

The current study aims to evaluate the effectiveness of predominantly self-help ACT interventions (web-based and bibliotherapy programs) in comparison to an education intervention among adults living with chronic pain.

The current study was a randomized controlled trial (RCT) with two experimental groups and an active control group. The first experimental group received access to an internet platform with videos, interactive content and exercises based on ACT. The second experimental group received a copy of a self-help book based on ACT for chronic pain and had access to this book's website which includes audio mindfulness exercises. The third group consisted of an active control group, in which participants received pamphlet style pdf documents of education for pain (without any ACT components) as well as related practical exercises.

DETAILED DESCRIPTION:
This study aimed to evaluate the effectiveness of a web-based ACT intervention program with minimal therapeutic contact, compared to an ACT-based bibliotherapy and a pain education program (active control group) among adults with chronic pain. Participants were randomly assigned to each group. We hypothesized that:

1. both ACT interventions would lead to significant reductions in pain-related disability (primary variable), greater than the control group (education), and that the web-based program would lead to greater reductions in disability than the bibliotherapy group;
2. both ACT interventions would lead to significant improvements in quality of life (secondary variable), greater than the control group (education), and that the web-based program would lead to greater improvements in quality of life than the bibliotherapy group;
3. both ACT interventions would lead to significant reductions in anxiety and depressive symptoms (secondary variables), greater than the control group (education), and that the web-based program would lead to greater reductions in anxiety and depressive symptoms than the bibliotherapy group;
4. Improvements on primary (pain-related disability) and secondary variables (quality of life, anxiety/depressive symptoms) for the ACT groups will be maintained at 3 and 6 months and will remain superior to the control group (education);
5. Participants from both ACT groups would have a positive impressions of change following the intervention (as measured by the PGIC scale).

   * Some of the questionnaires described in the following section were administered and will be subject to subsequent analyses examining patient trajectories of change and profiles of patients who respond well or not to these treatment modalities.

ELIGIBILITY:
Inclusion criteria:

1. Being 18 years or older;
2. Residing in Canada;
3. Having daily pain for at least 6 months;
4. Having a reading and writing ability equivalent or superior to grade 8;
5. Having access to internet at home and a valid e-mail address;
6. Not having previously engaged in an ACT-based psychotherapy and/or regularly meditated and/or read "Libérez-vous de la douleur" by Frédérick Dionne;
7. Not being in an unstable psychological situation (severe suicidal thoughts or severe/persistent mental health disorder);
8. Having an average level of pain of at least 4/10 within the past week;
9. Having non-cancer related pain;
10. Having stable medication for at least one month.

Participants were excluded if they did not meet any of the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Pain interference | Change from week start of treatment (week 0) to end of treatment (week 9), 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The Brief Pain Inventory (BPI) evaluates the severity and interference of pain in daily activities (Cleeland & Ryan, 1994; Tyler et al., 2002; French version: Poundja et al., 2007). The instrument consists of 10 items rated on a Likert scale ranging from 0 = does not interfere to 10 = interferes completely, and participants are asked to rate the degree to which pain interfered with various activities in the past week (e.g., social activities, work, mood, etc.). Higher scores represent higher levels of pain interference. This questionnaire has shown good reliability across a variety of populations (e.g. French speaking fibromyalgia patients; Bourgault et al., 2015). The BPI is extensively used in chronic pain research, has strong psychometric properties and is recommended as an outcome in clinical trials of patients with chronic pain (Dworkin et al., 2005). The French version has shown to have good internal consistency (Poundja et al., 2007).

SECONDARY OUTCOMES:
Change in Anxiety and Depression symptoms | Change from week start of treatment (week 0) to end of treatment (week 9), 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The Hospital Anxiety Depression Scale (HADS; Zigmond & Snaith, 1983; French version: Bocéréan & Dupret, 2014) is a 14-item questionnaire which evaluates psychological distress according to two 7-item subscales measuring anxiety and depressive symptoms in non-psychiatric hospital contexts. Items are scored on a 4-point Likert scale ranging from 0 to 3. An example of items is "I feel tense or wound up". A higher score reflects a higher level of anxiety or depression.
Change in Quality of life measure | Change from week start of treatment (week 0) to end of treatment (week 9), 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The World Health Organization Quality of Life-Brief (WHOQOL-BRIEF; WHOQOL; Group, 1998) is a self-reported measure of 26 items assessing quality of life in terms of physical and psychological health, social relationships and social functioning. Items are rated from 1 = very poor to 5 = very good, with higher scores reflect higher quality of life. This instrument has demonstrated good levels of internal consistency for its subscales (α = .66 to α = .80) and adequate test-retest reliability (r = .75). The French version of the instrument offers high internal consistency (Baumann, Erpelding, Régat, Collin, & Briançon, 2010).

OTHER OUTCOMES:
Psychological In/Flexibility | Change from week start of treatment (week 0) to end of treatment (week 9), 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The Multidimensional Psychological Flexibility Inventory (MPFI; Rolffs, Rogge & Wilson, 2016) is a 24 item scale that measures psychological flexibility and inflexibility processes. Items are rated on a six-point Likert scale ranging from 1 = never true to 6 = always true. This tool provides 12 distinct dimensions of flexibility or psychological influence.
Chronic Pain Acceptance | Change from week start of treatment (week 0) to end of treatment (week 9), 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The Chronic Pain Acceptance Questionnaire (CPAQ-8; Fish et al., 2010; Scott et al., 2013 ) is an 8-item version of the Chronic Pain Acceptance Questionnaire (McCracken et al., 2004). This measure is comprised of two subscales: activity engagement and pain willingness. Specific items include, "I am getting on with the business of living no matter what my level of pain is" and "Keeping my pain level under control takes first priority whenever I am doing something". Items are scored on a 7-point Likert scale ranging from 0 = never true to 6 = always true. Scores for the pain willingness subscale are reversed before calculating a total score so that higher total scores reflect greater levels of pain acceptance. The CPAQ has been used frequently in research and the short version has good psychometric properties (Fish et al., 2010).
Chronic Pain Self-Efficacy | Change from week start of treatment (week 0) to end of treatment (week 9), 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The French-Canadian Chronic Pain Self-Efficacy Scale (Lacasse et al., 2015; Lorig et al., 1996) is a 6-item scale that measures an individual's confidence in his/her ability to manage chronic pain in general and pain-related symptoms. Items are rated on a 10-point Likert scale ranging from 1 = not at all confident to 10 = entirely confident. A higher score reflects greater chronic pain self-efficacy. This scale has good psychometric properties (Lacasse et al., 2015).
Patient's Impression of Change | 3-month follow-up (week 22) and 6-month follow-up (week 35)
  The Patient Global Impression of Change (PGIC; Guy, 1976) is a 5-item tool evaluates the level of change perceived by the participant regarding his/her pain, physical functioning, quality of life and psychological well-being over the last three months.25 The statements are evaluated according to a 7-point Likert scale (e.g.: "Over the last 3 months, your functioning 0) has deteriorated considerably; 3) has remain unchanged or 6) has improved considerably"). A fifth item evaluates pain relief over the last 3 months and is measured according to an ordinal scale ranging from 0 (no relief) to 100 (total relief). Although it is widely used in clinical trials on CP, the validity of this scale has not been officially evaluated (Ferguson & Scheman, 2009) but its use is indicated by the IMMPACT expert group.
Diary items | Weekly changes from baseline (week 0), throughout treatment (Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9), and after treatment (week 10)
  In addition to pretreatment, posttreatment, and three and six-month follow-up assessments, participants were asked to answer 7 items assessing the three main axis of the ACT psychological flexibility model ("open", "aware" and "active"; Hayes et al., 2011) as well as four outcome variables (pain-related disability, anxiety, depression, and quality of life). The three items assessing ACT processes have been used in previous research (Scott et al., 2017) and were translated in French and slightly modified for the present study. More specifically, the original English version of items refers to the last three days, whereas we modified the questions to refer to the past seven days since measures were intended to be completed weekly. All items were rated on a Likert scale ranging from 0 (Never) to 6 (Always).

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Dionne, Ph.D., Study Director — Université du Québec à Trois-Rivières; Marie-Eve Martel, Psy.D., Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03711851/Prot_SAP_000.pdf